CLINICAL TRIAL: NCT00709488
Title: A Phase 1 Study to Evaluate the Safety and Effectiveness of Using the Litx™ BPH System in Patients With Lower Urinary Tract Symptoms (LUTS) Due to Benign Prostatic Hyperplasia (BPH) Who Are Candidates for Interventional Therapy
Brief Title: Phase 1 Study of the Litx™ BPH System in Patients With Lower Urinary Tract Symptoms (LUTS) Due to Benign Prostatic Hyperplasia (BPH)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Light Sciences Oncology (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LSO-OL008
Record Dates: First submitted 2008-06-30; First posted 2008-07-03 (Estimated); Last update posted 2012-11-16 (Estimated); Status verified 2012-11

CONDITIONS: Benign Prostatic Hyperplasia; Lower Urinary Tract Symptoms
Keywords: Litx™ BPH System; LS11; Talaporfin sodium
MeSH Terms: conditions — Prostatic Hyperplasia; Lower Urinary Tract Symptoms | interventions — Talaporfin; Embryo Implantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Litx™ BPH Therapy (Experimental)
  Interventions: Drug: Talaporfin sodium; Procedure: Placement of device in prostate urethra; Device: Transurethral illumination with light emitting diodes (Litx™ BPH Device)

INTERVENTIONS:
Drug: Talaporfin sodium — LS11 (Talaporfin Sodium) dose is 1mg/kg administered intravenously slow push (3-5 minutes).
  Other Names: LS11; Mono-L-aspartyl Chlorin e6
Procedure: Placement of device in prostate urethra — Placement of device in prostate urethra
Device: Transurethral illumination with light emitting diodes (Litx™ BPH Device) — Patients in Cohort A will receive 50 J of light treatment with 1 mg/kg LS11 administration; patients in Cohort B will receive 70 J of light treatment with 1 mg/kg LS11 administration; patients in Cohort C will receive 100 J of light treatment with 1 mg/kg LS11 administration; patients in Cohort D will receive 100 J of light treatment (with the active light emitting length increased from 10mm to 20 mm) with 1 mg/kg LS11 administration.

SUMMARY:
This is a phase 1 study to evaluate the safety and effectiveness of using the Litx™ BPH System in patients with LUTS due to benign prostatic hyperplasia (BPH).

DETAILED DESCRIPTION:
The eligible patients will be enrolled into one of the three Litx™ treatment Cohorts (A, B or C)

All patients will undergo the procedure of Litx™ BPH Device placement into the prostate urethra.

Following the placement of the Litx™ BPH Device into the urethra, patients in Cohort A will be administered an intravenous dose of LS11 (talaporfin sodium) at 1 mg/kg by slow push over 3 - 5 minutes. Fifteen minutes after injection, each patient will be administered a 50 J total light dose, delivered at 20 mW/cm over a 42 minute time period.

Following the placement of the Litx™ BPH Device into the urethra, patients in Cohort B will receive LS11 intravenously at 1 mg/kg by slow push over 3 to 5 minutes. The light activation procedure is the same as that for Cohort A except that a light dose of 70 J will be delivered to each patient over a 58 minute time period.

Following the placement of the Litx™ BPH Device into the urethra, patients in Cohort C will receive LS11 intravenously at 1 mg/kg by slow push over 3 to 5 minutes. The light activation procedure is the same as that for Cohort A except that a light dose of 100 J will be delivered to each patient over a 83 minute time period.

Following the placement of the Litx™ BPH Device into the urethra, patients in Cohort D will receive LS11 intravenously at 1 mg/kg by slow push over 3 to 5 minutes. The light activation procedure is the same as that for Cohort C except that the active light emitting length is 20 mm instead of 10mm.

After 30 days, patients who have not experienced an improvement in symptoms, as determined by the investigator, may undergo an additional interventional therapy with continued follow-up per the protocol.

Four weeks following treatment of the last patient in the current cohort, the number of patients requiring surgical intervention for relief of primary symptoms will be assessed for futility of the protocol prior to commencing with treatment of the first patient in the next consecutive cohort.

Upon acceptable safety assessment four weeks after completing the last patient treatment in each cohort, the first patient in the next consecutive cohort may be treated.

ELIGIBILITY:
Inclusion Criteria:

* Males, 50 years or older, who are on an alpha blocker and/or a 5-alpha reductase inhibitor or a combination, and are candidates for interventional therapy. Patients to continue on an alpha blocker and/or 5-alpha reductase inhibitor for at least one-month after the Litx™ treatment, then tapered off medication at physician's discretion.
* Patients who understand and have the ability to sign written informed consent prior to any study procedures and discontinuation of exclusionary medications.
* Patients with moderate to severe BPH bother score >3 requiring non-medication intervention.
* Patients with an IPSS1 Score of >15 points.
* Maximum urinary flow rate (Qmax) ≤15 mL/sec.
* Post void residual volume (PVR) ≤300 mL.
* Prostatic volume >50g by TRUS.

Exclusion Criteria:

* Patients with any previous minimally invasive or surgical intervention for BPH.
* Patients who have enrolled, or are currently enrolled in, another clinical trial for any disease within the past 30 days.
* Patients with an active urinary tract infection.
* Patients with a urethral stricture.
* Patients with a predominant middle lobe obstruction.
* Patients who have evidence or history of prostate or bladder cancer.
* Patients with a PSA of >10 ng/ml. If the PSA is 4-10 ng/ml, preliminary biopsy should be done within one-year prior to entry into the study to rule out prostate cancer.
* Patients who had a biopsy of the prostate within the past 6 weeks.
* Patients with bleeding diathesis.
* Patients with clinically significant renal or hepatic impairment.
* Patients with neurological conditions felt to affect the bladder or a history of a neurogenic or chronically decompensated bladder.
* Patients who daily use a pad or device for incontinence.
* Patients who had an episode of unstable angina pectoris, myocardial infarction, transient ischemic attack, or cerebrovascular accident (stroke) within the past 6 months, or peripheral arterial disease with intermittent claudication or Leriches syndrome.
* Patient has an interest in future fertility.
* Patients with prolonged QT interval at baseline or currently taking medications that prolong QT interval (prolonged QT interval defined as > 450 ms).
* Inadequate organ function as evidenced by the following: Platelet count <100,000/mm³; WBC <4,000/mm³; Neutrophils <1,800/mm³; Hemoglobin <10 g/dL; SGOT and SGPT >3 x ULN; Creatinine >1.2 mg/dL
* Known sensitivity to porphyrin-type drugs or known history of porphyria.
* Known sensitivity to antibiotics (i.e., levofloxacin, gentamicin, etc.).
* Inability to avoid sunlight after procedure during the first 2 weeks after LS11 administration.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2008-06; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Safety of Litx™ BPH System by Recording of Adverse Events; Preliminary effectiveness of Litx™ BPH System by evaluating the International Prostate Symptom Score (IPSS) along with Bother Score (BS). | 9 months

SECONDARY OUTCOMES:
To assess the effect of the Litx™ treatment following tests by: Maximum urinary flow rate (Qmax); Post void residual volume (PVR); Transrectal ultrasound (TRUS) to measure prostate size and treatment effect. | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Sy-Shi Wang, PhD, Study Director — Light Sciences Oncology, Inc
Locations (6):
- United States (6):
  - Alaska Clinical Research Center, Anchorage, Alaska
  - UCLA School of Medicine, GU Clinical Trials Office, Los Angeles, California
  - The Portland Clinic, Portland, Oregon
  - Urology San Antonio Research, San Antonio, Texas
  - Integrity Medical Research, Mountlake Terrace, Washington
  - Seattle Urological Associates, Seattle, Washington